CLINICAL TRIAL: NCT03244475
Title: Passive Electrical Neurofeedback Treatment of mTBI: MEG and Behavioral Outcomes
Brief Title: Transcranial Electrical Stimulation for mTBI
Acronym: TESmTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1988-I; RX001988-01A1 (Other Grant/Funding Number: Office of Research and Development)
Record Dates: First submitted 2017-07-24; First posted 2017-08-09 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Mild Traumatic Brain Injury (mTBI); Post-traumatic Stress Disorder
Keywords: mild Traumatic Brain Injury; transcranial electrical stimulation; neurofeedback; magnetoencephalography; post-traumatic stress disorder
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: After consent, Visit 1 (V1) for all 3 groups will include baseline NP and MHA. Then, baseline rs-MEG and MRI will be performed in V2 for all groups. At V3 the mTBI Veterans in TES and sham groups will undergo a pre-session MEG, the first TES/Sham treatment Session (S1), and a post-session MEG. Next, the mTBI Veterans continue their TES/Sham treatments S2-6 in V4-8. During V9, a pair of pre- and post-MEG exams and NP will be performed. The mTBI Veterans will continue treatments S8-11 in V10-13. During V14, a pair of pre- and post-MEG exams will be performed. 1 week after the Veterans finish their final TES/Sham treatment S12, a 1-week follow-up MEG and NP will be conducted during V15. A subset of TES group will be tested 1 month after the final treatment for a follow-up MEG V16. Veterans in the mTBI-sham group will be offered the real TES treatment.
Who Masked: Participant, Care Provider
Masking Description: Sham treatment, double-blind design: During the sham treatment, we will prep and preplace the electrodes for common reference, A-, B-, plus the set of electrodes on the scalp of the participant following the 10-20 EEG configuration for A+ and A-, just like the procedure for real TES treatment. However, no LIP-tES pulses will be sent from the system during sham treatment, based a code entered to the system. A staff member (SRA #1) will assign a mTBI Veteran to either the mTBI-TES or the mTBI Sham group, with an attached code from an existing code bank. Then, the TES treatment operator (SRA #2) who is blind to the group assignment will enter the code to the TES system during treatments. Based on the code, the system automatically loads the protocol for either TES or Sham treatment. Only at the end of the study (after V16), the group assignment is revealed. Therefore, both the participant and TES treatment operator (SRA #2) are blind to the group assignment during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Transcranial Electrical Stimulation (TES) (Experimental): mTBI Veterans blindly assigned to a 6 week of TES, either IASIS neurofeedback treatment or Nexalin, with 2-3 sessions per week.
  Interventions: Device: TES
- Sham Treatment (Placebo Comparator): mTBI Veterans blindly assigned to a sham treatment for 6 weeks with 2-3 sessions per week.
  Interventions: Device: TES
- Control (No Intervention): Veterans who are age-, gender-, education-, combat exposure-, and socioeconomically-matched. They will not undergo a treatment.

INTERVENTIONS:
Device: TES — The EEG interface device is the J&J Engineering I-330 C2. IASIS is delivered via the 4 EEG leads with respect to the Common Neck Reference. During each session, 2 electrodes are attached to the participant's left and right mastoids, while the remaining 2 electrodes are moved to various locations on the scalp to record EEG signals. All 4 electrodes are involved in applying weak electric current pulses back to the brain. The feedback signal consists 2 types of narrow pulse trains, both with 150mV in amplitude.
  The Nexalin device, FDA clearance (501K=K024377, Classification: Stimulator, Cranial Electrotherapy: CFR 882. 5800: U.S. Patent #6904322B2), produces a waveform that provides tES to the brain delivered at a frequency of 4Hz, 40Hz, and 77.5Hz at 0 to 15mA peak current. Evidence shows this waveform, at these frequencies, results in improved clinical outcomes for anxiety and pain. We hypothesize that repeated TES treatments serve to stimulate long-term neurochemical changes.
  Other Names: LIP-tES intervention
  Arms: Sham Treatment; Transcranial Electrical Stimulation (TES)

SUMMARY:
mTBI is a leading cause of sustained physical, cognitive, emotional, and behavioral deficits in OEF/OIF/OND Veterans and the general public. However, the underlying pathophysiology is not completely understood, and there are few effective treatments for post-concussive symptoms (PCS). In addition, there are substantial overlaps between PCS and PTSD symptoms in mTBI. IASIS is among a class of passive neurofeedback treatments that combine low-intensity pulses for transcranial electrical stimulation (LIP-tES) with EEG monitoring. Nexalin is another tES technique , with FDA approvals for treating insomnia, depression, and anxiety. LIP-tES techniques have shown promising results in alleviating PCS individuals with TBI. However, the neural mechanisms underlying the effects of LIP-tES treatment in TBI are unknown, owing to the dearth of neuroimaging investigations of this therapeutic intervention. Conventional neuroimaging techniques such as MRI and CT have limited sensitivity in detecting physiological abnormalities caused by mTBI, or in assessing the efficacy of mTBI treatments. In acute and chronic phases, CT and MRI are typically negative even in mTBI patients with persistent PCS. In contrast, evidence is mounting in support of resting-state magnetoencephalography (rs-MEG) slow-wave source imaging (delta-band, 1-4 Hz) as a marker for neuronal abnormalities in mTBI. The primary goal of the present application is to use rs-MEG to identify the neural underpinnings of behavioral changes associated with IASIS treatment in Veterans with mTBI. Using a double-blind placebo controlled design, the investigators will study changes in abnormal MEG slow-waves before and after IASIS treatment (relative to a 'sham' treatment group) in Veterans with mTBI. For a subset of participants who may have remaining TBI symptoms at the end of all IASIS treatment sessions, MEG slow-wave changes will be recorded before and after additional Nexalin treatment. In addition, the investigators will examine treatment-related changes in PCS, PTSD symptoms, neuropsychological test performances, and their association with changes in MEG slow-waves. The investigators for the first time will address a fundamental question about the mechanism of slow-waves in brain injury, namely whether slow-wave generation in wakefulness is merely a negative consequence of neuronal injury or if it is a signature of ongoing neuronal rearrangement and healing that occurs at the site of the injury.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI) is a leading cause of sustained physical, cognitive, emotional, and behavioral deficits in OEF/OIF/OND Veterans and the general public. However, the underlying pathophysiology is not completely understood, and there are few effective treatments for post-concussive symptoms (PCS). In addition, there are substantial overlaps between PCS and post-traumatic stress disorder (PTSD) symptoms in mTBI. Furthermore, a substantial number of studies have shown higher (nearly double) rates of comorbid PTSD in individuals with mTBI, observed in military and civilian settings. IASIS is among a class of passive neurofeedback treatments that combine low-intensity pulses for transcranial electrical stimulation (LIP-tES) with electroencephalography (EEG) monitoring. Nexalin is another tES technique , with FDA approvals for treating insomnia, depression, and anxiety. LIP-tES techniques have shown promising results in alleviating PCS in individuals with TBI. However, the neural mechanisms underlying the effects of LIP-tES treatment in TBI are unknown, owing to the dearth of neuroimaging investigations of this therapeutic intervention. Conventional neuroimaging techniques such as MRI and CT have limited sensitivity in detecting physiological abnormalities caused by mTBI, or in assessing the efficacy of mTBI treatments. In acute and chronic phases, CT and MRI are typically negative even in mTBI patients with persistent PCS. In contrast, evidence is mounting in support of resting-state magnetoencephalography (rs-MEG) slow-wave source imaging as a non-invasive imaging marker for neuronal abnormalities in mTBI. Using region of interest (ROI) and voxel-wise approaches, the investigators demonstrated that MEG slowwave source imaging detects abnormal slow-waves (delta-band, 1-4 Hz) with ~85% sensitivity in chronic and sub-acute mTBI patients with persistent PCS. The primary goal of the present application is to use rs- MEG to identify the neural underpinnings of behavioral changes associated with IASIS treatment in Veterans with mTBI. Using a double-blind placebo controlled design, the investigators will study changes in abnormal MEG slowwaves before and after IASIS treatment (relative to a 'sham' treatment group), and for a subset, before and after additional Nexalin treatment, in Veterans with mTBI. In addition, the investigators will examine treatment-related changes in PCS, PTSD symptoms, neuropsychological test performances, and their association with changes in MEG slow-waves. Pre-treatment baseline and posttreatment rs-MEG exams, symptoms assessments, and neuropsychological tests will be performed. The investigators for the first time will address a fundamental question about the mechanism of slow-waves in brain injury, namely whether slow-wave generation in wakefulness is merely a negative consequence of neuronal injury or if it is a signature of ongoing neuronal rearrangement and healing that occurs at the site of the injury.

Specific Aim 1: To detect the loci of injury in Veterans with mTBI and assess the mechanisms underlying functional neuroimaging changes related to IASIS treatment, and for a subset of Veterans with remaining symptoms, additional Nexalin treatment, using rs-MEG slow-wave source imaging. The investigators' voxel-wise rs-MEG source-imaging technique will be used to identify abnormal slow-wave generation (delta band) in the baseline and post-treatment MEG exams to assess treatment-related changes on a single-subject basis. Healthy control (HC) Veterans, matched for combat exposure, will be used to establish an MEG normative database. Test-retest reliability of MEG slow-wave source imaging for mTBI will also be examined.

Hypothesis 1: Veterans with mTBI will generate abnormal MEG slow-waves during the baseline MEG exam. Voxel-wise MEG slow-wave source imaging will show significantly higher sensitivity than conventional MRI in identifying the loci of injury on a single-subject basis. The test-retest reliability of MEG slow-wave source imaging is expected to be high, with intra-class correlation coefficient (ICC) 0.75 between two sequential MEG exams.

Hypothesis 2: In wakefulness, slow-wave generation is a signature of ongoing neural rearrangement/ healing, rather than a negative consequence of neuronal injury. IASIS treatment will enhance neural rearrangement/healing by initially potentiating slow-wave generation immediately after each treatment session.

Hypothesis 3: IASIS will ultimately reduce abnormal MEG slow-wave generation in mTBI by the end of the treatment course, owing to the accomplishment of neural rearrangement / healing. In Veterans with mTBI who finish IASIS treatment, but not in the sham group, MEG source imaging will show a significant decrease in abnormal slow-waves at post-treatment exam. Such significant decreases will also be evident in both the voxel-wise and overall abnormal MEG slow-wave measures.

Specific Aim 2: To examine treatment-related changes in PCS and PTSD symptoms in Veterans with mTBI. PCS and PTSD symptoms will be assessed at the baseline and post-treatment follow-up visits.

Hypothesis 4: Compared with the sham group, mTBI Veterans in the IASIS treatment group will show significantly greater decreases in PCS symptoms between baseline and post-treatment assessments.

Hypothesis 5: Compared with the sham group, mTBI Veterans in the IASIS treatment group will also show significantly greater decreases in PTSD symptoms between baseline and post-treatment assessments.

Specific Aim 3: To study the relationship among IASIS treatment-related changes in rs-MEG slow-wave imaging, PCS, and neuropsychological measures in Veterans with mTBI. The investigators will correlate changes between baseline and post-IASIS abnormal rs-MEG slow-wave generation (i.e., total abnormal rs-MEG slow-wave and voxel-wise source imaging measures) with changes in PCS and neuropsychological tests performance.

Hypothesis 6: Reduced MEG slow-wave generation will correlate with reduced total PCS score, individual PCS scores (e.g., sleep disturbance, post-traumatic headache, photophobia, and memory problem symptoms), and improved neuropsychological exam scores between post-IASIS and baseline exams.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of Veterans for the mTBI groups:

* All symptomatic mTBI patients will be evaluated in a clinical interview to document the nature of the injuries and ongoing PCS.
* The diagnosis of mTBI patients is based on standard VA/DOD diagnostic criteria.
* Inclusion in the mTBI patient group requires a TBI that meets the following criteria:

  * a loss of consciousness (LOC) < 30 minutes or transient confusion, disorientation, or impaired consciousness immediately after the trauma
  * post-traumatic amnesia (PTA) < 24 hours
  * an initial Glasgow Coma Scale (GCS) [90] between 13-15 (if available)
* Since the GCS assessment is often not available in theater, Veterans with missing GCS, but who meet other inclusion criteria will also be recruited.
* Each patient must have at least 3 items of persistent PCS at the beginning of the study.

Inclusion of Healthy Control (HC) group:

* Veterans that qualify as HCs will be age, education, combat exposure, and socioeconomically matched to the mTBI groups.
* In addition to exclusion criteria listed above, HC subjects must not have been diagnosed with head injury, affective disorder, or PTSD (CAPS-5 < 8) throughout life.

Exclusion Criteria:

* Exclusion criteria for study participations include:
* history of other neurological, developmental, or psychiatric disorders (based on the DSM-5 (MINI-7) [86] structured interview), e.g.,:

  * brain tumor
  * stroke
  * epilepsy
  * Alzheimer's disease
  * schizophrenia
  * bipolar disorder
  * ADHD
  * or other chronic neurovascular diseases such as hypertension and diabetes
* substance or alcohol use disorders according to DSM-5 [87] criteria within the six months prior to the study
* history of metabolic or other diseases known to affect the central nervous system (see [88] for similar criteria)
* Metal objects (e.g., shrapnel or metal fragments) that fail MRI screening, or extensive metal dental hardware, e.g.,:

  * braces and large metal dentures

    * fillings are acceptable
  * other metal objects in the head
  * neck, or face areas that cause non-removable artifacts in the MEG data
* Potential subjects will be administered the Beck Depression Inventory (BDI-II) to evaluate level of depressive symptoms, and suicidal ideation

  * any participant who reports a "2" or "3" on the BDI-II: item 9 (suicidal thoughts or wishes) will also be excluded.
  * However, depression following mTBI or traumatic event of PTSD is common [89]: therefore, in two mTBI groups, the investigators will include and match patients with depression symptoms reported after their injury/event, and will co-vary BDI-II score in data analyses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingxiong Huang, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
One or more data sets without personal identifiers will be generated during the data analysis phase of this study. Publications from this research will be made available to the public through the National Library of Medicine PubMed Central website within one year after the date of publication. The data sets will include all data underlying any publications generated by this study and therefore, these will be sufficient to reproduce or verify any published findings.
  Requests for access to final data sets must be made in writing signed by a requestor from the United States and include an email address for delivery and an assurance that the recipient will not attempt to identify or re-identify any individual. The request should reference the publication underlying the request. Requests may be made to the PI/lead point-of-contact for the publication. If the investigator leaves the VASDHS the requests may be sent to the Associate Chief of Staff for Research.

REFERENCES:
- [Background] Huang MX, Nichols S, Baker DG, Robb A, Angeles A, Yurgil KA, Drake A, Levy M, Song T, McLay R, Theilmann RJ, Diwakar M, Risbrough VB, Ji Z, Huang CW, Chang DG, Harrington DL, Muzzatti L, Canive JM, Christopher Edgar J, Chen YH, Lee RR. Single-subject-based whole-brain MEG slow-wave imaging approach for detecting abnormality in patients with mild traumatic brain injury. Neuroimage Clin. 2014 Jun 16;5:109-19. doi: 10.1016/j.nicl.2014.06.004. eCollection 2014. PMID 25009772
- [Background] Huang M, Risling M, Baker DG. The role of biomarkers and MEG-based imaging markers in the diagnosis of post-traumatic stress disorder and blast-induced mild traumatic brain injury. Psychoneuroendocrinology. 2016 Jan;63:398-409. doi: 10.1016/j.psyneuen.2015.02.008. Epub 2015 Feb 23. PMID 25769625
- [Background] Robb Swan A, Nichols S, Drake A, Angeles A, Diwakar M, Song T, Lee RR, Huang MX. Magnetoencephalography Slow-Wave Detection in Patients with Mild Traumatic Brain Injury and Ongoing Symptoms Correlated with Long-Term Neuropsychological Outcome. J Neurotrauma. 2015 Oct 1;32(19):1510-21. doi: 10.1089/neu.2014.3654. Epub 2015 Jun 18. PMID 25808909
- [Background] MacGregor AJ, Dougherty AL, Galarneau MR. Injury-specific correlates of combat-related traumatic brain injury in Operation Iraqi Freedom. J Head Trauma Rehabil. 2011 Jul-Aug;26(4):312-8. doi: 10.1097/HTR.0b013e3181e94404. PMID 20808241
- [Background] MacDonald CL, Johnson AM, Nelson EC, Werner NJ, Fang R, Flaherty SF, Brody DL. Functional status after blast-plus-impact complex concussive traumatic brain injury in evacuated United States military personnel. J Neurotrauma. 2014 May 15;31(10):889-98. doi: 10.1089/neu.2013.3173. Epub 2014 Feb 10. PMID 24367929
- [Background] Hoffman SW, Harrison C. The interaction between psychological health and traumatic brain injury: a neuroscience perspective. Clin Neuropsychol. 2009 Nov;23(8):1400-15. doi: 10.1080/13854040903369433. PMID 19882478
- [Background] Vasterling JJ, Brailey K, Proctor SP, Kane R, Heeren T, Franz M. Neuropsychological outcomes of mild traumatic brain injury, post-traumatic stress disorder and depression in Iraq-deployed US Army soldiers. Br J Psychiatry. 2012 Sep;201(3):186-92. doi: 10.1192/bjp.bp.111.096461. Epub 2012 Jun 28. PMID 22743844
- [Background] Nelson DV, Esty ML. Neurotherapy of Traumatic Brain Injury/Post-Traumatic Stress Symptoms in Vietnam Veterans. Mil Med. 2015 Oct;180(10):e1111-4. doi: 10.7205/MILMED-D-14-00696. PMID 26444476
- [Background] Schoenberger NE, Shif SC, Esty ML, Ochs L, Matheis RJ. Flexyx Neurotherapy System in the treatment of traumatic brain injury: an initial evaluation. J Head Trauma Rehabil. 2001 Jun;16(3):260-74. doi: 10.1097/00001199-200106000-00005. PMID 11346448
- [Background] Huang MX, Nichols S, Robb A, Angeles A, Drake A, Holland M, Asmussen S, D'Andrea J, Chun W, Levy M, Cui L, Song T, Baker DG, Hammer P, McLay R, Theilmann RJ, Coimbra R, Diwakar M, Boyd C, Neff J, Liu TT, Webb-Murphy J, Farinpour R, Cheung C, Harrington DL, Heister D, Lee RR. An automatic MEG low-frequency source imaging approach for detecting injuries in mild and moderate TBI patients with blast and non-blast causes. Neuroimage. 2012 Jul 16;61(4):1067-82. doi: 10.1016/j.neuroimage.2012.04.029. Epub 2012 Apr 20. PMID 22542638
- [Background] Huang MX, Theilmann RJ, Robb A, Angeles A, Nichols S, Drake A, D'Andrea J, Levy M, Holland M, Song T, Ge S, Hwang E, Yoo K, Cui L, Baker DG, Trauner D, Coimbra R, Lee RR. Integrated imaging approach with MEG and DTI to detect mild traumatic brain injury in military and civilian patients. J Neurotrauma. 2009 Aug;26(8):1213-26. doi: 10.1089/neu.2008.0672. PMID 19385722
- [Background] Lewine JD, Davis JT, Bigler ED, Thoma R, Hill D, Funke M, Sloan JH, Hall S, Orrison WW. Objective documentation of traumatic brain injury subsequent to mild head trauma: multimodal brain imaging with MEG, SPECT, and MRI. J Head Trauma Rehabil. 2007 May-Jun;22(3):141-55. doi: 10.1097/01.HTR.0000271115.29954.27. PMID 17510590
- [Background] Lewine JD, Davis JT, Sloan JH, Kodituwakku PW, Orrison WW Jr. Neuromagnetic assessment of pathophysiologic brain activity induced by minor head trauma. AJNR Am J Neuroradiol. 1999 May;20(5):857-66. PMID 10369357

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Electrical Stimulation (TES): mTBI Veterans blindly assigned to a 6-week IASIS neurofeedback treatment with two sessions per week.
  If participants in the mTBI group may have remaining PCS, additional Nexalin treatment will be offered. Nexalin TES will be administered once per day, Monday through Friday. Participants will receive 10-20 treatments, 3-4 times a week for 4 weeks, or up to 5 times a week for 4 weeks.
- TES Sham Treatment: mTBI Veterans blindly assigned to a sham treatment for 6 weeks with two IASIS sessions per week or 10-20 Nexalin treatments, 3-4 times a week for 4 weeks or up to 5 times a week for 4 weeks.
Period: Overall Study
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Started | 30 | 17 | 19
Completed | 18 | 4 | 19
Not Completed | 12 | 13 | 0

BASELINE CHARACTERISTICS:
Population: mTBI Veterans enrolled in a blinded study group. At the end of their study sessions, they were informed of their study group. If they were originally in a sham group, they had the option of receiving TES sessions. Questionnaires and MEG imaging continued if they chose to receive actual TES sessions. Therefore, the number of analysis TES population (n=38) is higher than the number of enrolled participants since some participants completed sham treatments and then opted for TES treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control | Total
Number analyzed (Participants) | 30 | 17 | 19 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 17 | 19 | 66
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.17857143 (10.06072126) | 38.375 (6.945097192) | 39.68421053 (7.643728985) | 38.68253968 (8.677329332)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 29 | 15 | 18 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 5 | 14
  Not Hispanic or Latino | 22 | 16 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 17 | 19 | 66
Handedness [Number; unit: Participants Right Handed] | 28 | 17 | 19 | 64
Education Level [Mean (Standard Deviation); unit: years] — Years of education collected via demographics forms:
  High School = 12 AA = 14 BA/BS = 16 MA/MS = 18 JD = 19 MD, DO, ND: 20 PhD = 21 MD, MD/PhD = 25
  years | 15.03703704 (3.024363802) | 14.8125 (1.911110606) | 15.94736842 (2.139200151) | 15.25806452 (2.558574981)

OUTCOME MEASURES:

1. Primary Outcome: Change in Abnormal Magnetoencephalography (MEG) Slow-Waves (1-4 Hz) Activity
Description: We will develop a voxel-wise whole brain MEG source imaging approach for detecting abnormal Magnetoencephalography (MEG) slow-waves (1-4 Hz) in mTBI Veterans. The unit of the abnormal MEG source activity was measured in pico Ampere-meter (or pA-m which is 10^(-12) A-m). Natural logarithm transformation (i.e., e-based) was used. So, the unit of the MEG source imaging was log(pA-m). The range of the voxel-wise MEG source activity scale is 0-10. High amplitude of the MEG source activity suggests more serious injury. In the present study, we measured the Difference score in MEG exam pre- vs post the transcranial electrical stimulation (TES) treatment. Our primary measure is the reduction of the abnormal MEG source activity for slow waves (1-4 Hz), defined as the MEG activity at the pre-TES exam minus that at the post-TES exam. So, the higher this difference score is, the better outcomes due to the TES treatment in reducing the abnormal MEG signal.
Time Frame: Baseline through end of treatment, an average of 6 weeks
Population: # of TES participants analyzed differs from the # of TES participants enrolled. mTBI veterans who were blindly placed in the TES Sham group had the option of completing TES sessions at the end of their original sessions. Therefore, some TES Sham participants opted to complete TES sessions, with questionnaires and pre-post MEG imaging.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 38 | 17 | 19
units on a scale | 1.8 (1.2) | 0.2 (1.4) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; The analysis was performed for the voxel-wise delta-band activity from the frontal pole and inferior frontal gyri. Spatial smoothing and logarithm transformation (e-based) were performed. Resting-state MEG activity differences between pre- and post-treatment measures were obtained as difference scores for TES and Sham separately. The null hypothesis was that there was no group difference in the pre- and post-treatment difference scores between TES and Sham groups; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.01, Wilcoxon (Mann-Whitney) — The corrected p-value of 0.01 was chosen after the standard cluster analysis for correcting family-wise error across different voxels; Wilcoxon test was chosen due to potential non-normal distribution for the difference scores; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [1.1 to 2.2]

2. Primary Outcome: Rivermead Post Concussion Symptom Questionnaire
Description: The Rivermead Post Concussion Symptom Questionnaire (RPQ) total score was used to assess change in post-concussion symptoms due to TES. Our focus in this analysis was the difference score in RPQ total score pre- vs post-treatment measures.
  The questionnaire has 16 items and uses scale of 0 - 4, with 0 as "not experienced at all" and 4 as "a severe problem." Value range: 0 - 64, where the higher scores mean a worse outcome.
  For this measure, we focused on the difference score: total score from prior to treatment minus total score from end of treatment. Therefore, the higher the difference score, the more positive change was observed.
Time Frame: Baseline through end of treatment, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 25 | 15 | 19
units on a scale | 11.1 (9.7) | 10.9 (11.2) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; Differences between pre- and post-treatment measures were obtained as difference scores for TES and Sham separately. The null hypothesis was that there was no group difference in the pre- and post-treatment difference scores between TES and Sham groups; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

3. Primary Outcome: Neurobehavioral Symptoms Inventory
Description: The Neurobehavioral Symptoms Inventory (NSI) total score was used to assess the changes of post-concussion symptoms due to TES. Our focus in this analysis was the difference score in NSI total score pre- vs post-treatment measures.
  The NSI has 22 items and uses a response scale of 0 - 4, with 0 as "none" and 4 as "very severe." Value range: 0 - 88, where the higher scores mean a worse outcome/more severe post-concussive symptoms.
  For this measure, we focused on the difference score: total score from prior to treatment minus total score from end of treatment. Therefore, the higher the difference score, the more positive change was observed.
Time Frame: Baseline through end of treatment, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 25 | 15 | 19
units on a scale | 12.3 (13.0) | 12.7 (10.7) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

4. Secondary Outcome: The McGill Pain Questionnaire (MGPQ)
Description: The McGill Pain Questionnaire (MGPQ) will evaluate the level of current pain, pain changes over time, and strength of pain, since pain is frequently co-morbid with mTBI.
  Category scores range from 1-2 through 1-6. Minimum score = 0. Maximum score = 78. The higher the pain score, the greater the pain.
  For this measure, we focused on the difference score: total score from prior to treatment minus total score from end of treatment. Therefore, the higher the difference score, the more positive change was observed.
Time Frame: Baseline through end of treatment, an average of 6 weeks
Population: Some participants did not complete the MGPQ and/or did not complete all study visits, therefore, no statistical analysis was completed on this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 19 | 10 | 10
units on a scale | 14.8 (16.9) | -5.1 (18.1) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

5. Secondary Outcome: Clinician-Administered PTSD Scale (CAPS-5)
Description: The CAPS-5 is a standard semi-structured interview used to assess PTSD diagnosis and severity. The primary traumatic event is elicited and will be used as the basis of assessing PTSD symptoms. The total symptom severity score is calculated by summing severity scores assessed in this 30-item questionnaire. PTSD diagnostic status will be assessed using the past month version of the CAPS-5A, in which total severity score of 33 or higher indicates full threshold PTSD. The past week version of the CAPS-5 will be given prior to treatment and at follow-up.
  Severity scores range on a response scale of 0-5, 0=absent, 5=extreme/incapacitating. CAPS-55 summary scores range from 0 to 80, with the higher scores indicating greater severity of PTSD symptoms.
  For this measure, we focused on the difference score: total score from prior to treatment minus total score from end of treatment. Therefore, the higher the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 22 | 11 | 16
units on a scale | 6.5 (13.4) | 4.2 (9.6) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

6. Secondary Outcome: Post-Concussion Check List (PCL-5)
Description: PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 uses a response scale of 0 - 4. 0 = "Not at all" to 4 = "Extremely." The total score can range from 0 - 80, with the higher the score corresponding to a higher level of distress to the very stressful experience. The difference between scores post-treatment and pre-treatment will analyzed in addition to the CAPS-5 (1 week version) outcomes. DSM-5 symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster, i.e., cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20); these subscale scores may be used in secondary analysis.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 26 | 15 | 19
units on a scale | 14.9 (15.9) | 12.1 (24.3) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the DIFFERENCE scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

7. Secondary Outcome: California Verbal Learning Test-2nd Edition - Free Recall Total Correct T-score
Description: We will use T-scores from verbal learning and retrospective memory (California Verbal Learning Test-2nd Edition). Alternate CVLT forms were used during the post-treatment session.
  T-score ranges from 5 to 95, where the higher the T-score, the better the outcome. The T-score indicates the number of standard deviations away from the mean, where 50 is the mean with a standard deviation of 10, and is age- and gender-corrected.
  Analysis was based on the difference score between pre-treatment and post-treatment Free Recall Total Correct T-score. The lower the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: CVLT Free Recall Total Correct t-score
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 27 | 15 | 19
CVLT Free Recall Total Correct t-score | -6.7 (9.8) | -2.8 (7.4) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the DIFFERENCE scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

8. Secondary Outcome: Wechsler Adult Intelligence Scale-4th Edition (WAIS-IV) Processing Speed Index
Description: We will use the sum of scaled scores from the WAIS-IV Symbol Search and Coding subtests to attain the Processing Speed Index.
  PSI ranged from 50 - 150, where the higher the score, the better the outcome. Analysis was based on the difference score between pre-treatment Processing Speed Index and post-treatment Processing Speed Index. The lower the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 27 | 15 | 19
units on a scale | -5.06 (10.53) | -11.48 (11.21) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

9. Secondary Outcome: Delis-Kaplan Executive Function System (DKEFS) - Trail Number/Letter Switching Scaled
Description: Throughout the study, we used DKEFS Verbal Fluency, Trail-Making, and Color-Word Interference subtests to assess executive functioning.
  Analysis was based on the DKEFS Trailmaking Number/Letter Switching scaled score. Scaled scores range from 1-19, where the higher the scaled score, the better the outcome.
  Analysis was based on the difference score between pre-treatment scaled score and the post-treatment scaled score. The lower the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 27 | 15 | 19
units on a scale | -0.77 (1.13) | -2.08 (2.03) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

10. Secondary Outcome: Connors Continuous Performance Task II (CPT-II) - Inattention Omissions T-Score
Description: The Connors Continuous Performance Task II (CPT-II) was included as a measure of attention and impulsivity.
  In this measure, converted T-scores represent the score of the individual relative to the population, who are of the same gender and same age group. A T-score of 50 represents the average for the comparison group. T-score ranges from under 40 (very good performance) to 65+ (markedly atypical). The higher the scores, the worse the performance.
  This analysis focused on the difference score between the Inattention Omissions T-score pre- and post-treatment. The higher the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: Inattention Omissions T-score
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 27 | 15 | 19
Inattention Omissions T-score | 5.71 (8.04) | -0.89 (10.02) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the DIFFERENCE scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

11. Secondary Outcome: Barratt Impulsivity Scale
Description: Impulsivity was also measured by Barratt Impulsivity Scale, a self-report questionnaire.
  This scale contains 30 items, with total scores that range from 30 - 120. The higher the score, the worse the outcome.
  Analysis was based on the difference score between pre- and post-treatment. The higher the difference score, the more positive change was observed.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 24 | 15 | 19
units on a scale | 7.6 (8.1) | 2.4 (10.8) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the DIFFERENCE scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

12. Secondary Outcome: Frontal Systems Behavior Scale
Description: Since frontal lobe areas are more prone to damage, the Frontal Systems Behavior Scale (FrSBe) will measure behavioral dysfunction associated with frontal subcortical impairment.
  FrSBe is a 46-item rating scale with three subscales: Apathy (14 items), Disinhibition (15 items), and Executive Function (17 items). Items are rated in a 5-point scale, where higher scores mean a worse outcome. The raw scores of these subscales were converted to T-scores, with range of 9 - >/= 140, where T-scores greater than 65 are considered clinically significant.
  For this measure, we focused on the difference score of the total T-score prior to treatment minus total score from end of treatment. Therefore, the higher the difference score, the more positive change was observed.
Time Frame: Baseline through end of treatment, an average of 6 weeks
Population: Some participants did not complete the FrSBe and/or did not complete all study visits, but analysis was completed on those who finished the FRsBe.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
Number analyzed (Participants) | 24 | 15 | 15
T-score | 9.1 (13.1) | 3.2 (17.2) | 0 (0)
Statistical Analysis 1: Comparison: Transcranial Electrical Stimulation (TES) vs TES Sham Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Statistical analysis was carried out for the difference scores to assess group differences between TES and Sham groups; p = 0.05, Wilcoxon (Mann-Whitney); Wilcoxon test was chosen due to potential non-normal distribution for the difference scores

ADVERSE EVENTS:
Time Frame: Time period for collection of adverse event data: pre-treatment collection (1 week - 1 month), treatment/sham collection (6 weeks), and post-treatment collection (1 week - 1 month)
Description: Out of 66 total participants, we had 30 originally in the TES category, 17 in Sham, and 19 as controls. But 8 in the Sham requested to do TES afterwards. Therefore, we ended up with 38 TES overall.
Groups:
- Transcranial Electrical Stimulation (TES): mTBI Veterans blindly assigned to a 6-week IASIS or Nexalin TES treatment with two sessions per week.
  If participants in the mTBI group may have remaining PCS after IASIS, additional Nexalin TES treatment will be offered. Nexalin TES will be administered once per day, Monday through Friday. Participants will receive 10-20 treatments, 3-4 times a week for 4 weeks, or up to 5 times a week for 4 weeks.
  Out of 66 total participants, we had 30 originally in the TES category, 17 in Sham, and 19 as controls. But 8 in the Sham requested to do TES afterwards. So, we ended up with 38 TES overall.
Arm/Group | Transcranial Electrical Stimulation (TES) | TES Sham Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/38 | 0/17 | 0/19

LIMITATIONS AND CAVEATS:
Due to COVID restrictions and a long lock down period, this study was unable to enroll and consent Veteran participants for 7 months. Furthermore, some of the participants who enrolled pre-COVID were unable to complete all their treatment sessions nor their post-treatment MEG, neuropsychological testing, and mental health sessions. This has severely impacted data collection. We were able to start enrolling in October 2020. However, recruitment has been much slower than in the pre-COVID period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03244475/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT03244475/ICF_001.pdf